CLINICAL TRIAL: NCT01506089
Title: Optimizing the Temperature for Embryo Culture in In Vitro Fertilization: A Randomized Controlled Trial
Brief Title: Optimizing the Temperature for Embryo Culture in In Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RMA-2011-02
Record Dates: First submitted 2012-01-03; First posted 2012-01-09 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: IVF; infertility; PGD; embryo; temperature; incubator; CCS; culture; incubator-36 degrees Celsius; incubator-37 degrees Celsius
MeSH Terms: conditions — Infertility | interventions — Prostaglandins D; Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 36 degree group (Experimental): 36 degrees Celsius for the incubators is the experimental condition in this study.
  Interventions: Other: 36 degrees Celsius
- 37 degree group (No Intervention): 37 degrees Celsius is the standard incubator temperature for the culture of embryos.

INTERVENTIONS:
Other: 36 degrees Celsius — Embryos in this group will be cultured in incubators set to 36 degrees Celsius.
  Other Names: IVF, PGD, embryos, culture, CCS, infertility
  Arms: 36 degree group

SUMMARY:
Many human and animal studies over the past 40 years have revealed that ovaries and Fallopian tubes have a lower temperature than core body temperature, especially around the time of ovulation and early embryo development. Whether average core body temperature, 37 degrees Celsius, is ideal temperature for culture has not been prospectively evaluated. The purpose of this study is to determine whether lowering the incubator temperature by 1 degree Celsius will result in meaningful improvements in embryo development and pregnancy rates.

Patients participating in this study will undergo routine in vitro fertilization (IVF) stimulation. Following egg retrieval, patients with at least 8 mature eggs will have those eggs divided randomly into two groups. Both groups will then under ICSI (intra-cytoplasmic sperm injection) to fertilize the eggs. The groups will randomly be assigned to control or study condition. The control condition group will be cultured at 37 degrees Celsius, the current standard of care. The study group will be cultured at 36 degrees Celsius. All other culture conditions will be kept identical and embryos will be assessed on day 3 and day 5 of development.

On day 5, all well-developed blastocysts will undergo biopsy for Comprehensive Chromosomal Screening (CCS), which will evaluate the chromosomal normalcy of the embryo . Patients will undergo transfer on the morning of day 6 and the highest quality, chromosomally normal embryo from each group (the 36 degree cultured embryos and the 37 degree cultured embryos) will be transferred. If only 1 embryo is available for transfer, the patient will have a single embryo transfer.

All embryos available for cryopreservation will undergo biopsy for CCS before being frozen. Some arrested embryos from each temperature group will also undergo genetic analysis to evaluate chromosomal normalcy or mosaicism.

The female patient will undergo a blood draw at 9 weeks gestation and buccal swabs will be obtained from the infant(s) after birth.

ELIGIBILITY:
Inclusion Criteria:

* No more than 1 prior failed cycle at RMA NJ facility; up to 2 prior failed cycles at another facility pending investigator review
* Female partner between 18 and 41 at onset of IVF cycle
* Normal day 3 FSH (< or = 12) in RMA NJ laboratory
* Basal antral follicle count of at least 10
* Male partner with greater than 100,000 total motile spermatozoa per ejaculate (donor sperm is ok)
* BMI < or = 32 kg/m2

Exclusion Criteria:

* Diagnosis of chronic anovulation (cycles occuring typically less often than every 90 days)
* Use of testicular aspiration or biopsy procedures to obtain sperm
* Unevaluated ovarian mass or diagnosis of surgically-confirmed stage IV endometriosis
* Presence of hydrosalpinges that communicate with the uterine cavity
* History of endometrial insufficiency
* Any contraindication to undergoing IVF or gonadotropin stimulation
* Prior poor fertilization rate- less than 50% of mature eggs
* Prior poor blastulation rate- less than 10% of 2PNs (day 1 embryos)

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Useable Blastocyst Formation Rate | approximately 1 week
  Proportion of mature eggs developing into expanded blastocysts (Gardner grade 3-6) of sufficient quality to transfer or cryopreserve will be documented for each group (36 degree and 37 degree group).

SECONDARY OUTCOMES:
Fertilization rate | approximately 2 days
  The proportion of mature eggs that underwent ICSI and are normally fertlized (documented as forming 2 pro-nuclei (2PNs)) on the day after egg retrieval will be documented for each group (36 degree and 37 degree groups)
Cleavage Rate | approximately 1 week
  Proportion of properly fertlized embryo (2PNs on day 1) that undergo further celluar division will be documented for each group (36 degree and 37 degree group).
Blastocyst Formation Rate | approximately 1 week
  Proportion of mature oocytes that go on to develop into blastocysts in each group (36 degree group and 37 degree group) will be documented.
Implantation Rate | approximately 2 weeks
  Proportion of transferred embryos resulting in a clinically documented pregnancy will be documented for each group (36 degree and 37 degree group).
Aneuploidy Rate | approximately 1 month
  Rate of chromosomal abnormalities among the embryos in each group (36 degree and 37 degree groups) as determined by polymerase chain reaction (PCR) based comprehensive chromosome screening (CCS).
Mosaicism Rate | approximately 1 month
  Proportion of embryos that arrest at the cleavage stage which show evidence of more than one chromosomal lineages (mosaicism) when analyzed my microarray documented in each group (36 degree and 37 degree group).

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Associates of Pennsylvannia, Allentown, Pennsylvania

REFERENCES:
- [Derived] Hong KH, Lee H, Forman EJ, Upham KM, Scott RT Jr. Examining the temperature of embryo culture in in vitro fertilization: a randomized controlled trial comparing traditional core temperature (37 degrees C) to a more physiologic, cooler temperature (36 degrees C). Fertil Steril. 2014 Sep;102(3):767-73. doi: 10.1016/j.fertnstert.2014.06.009. Epub 2014 Jul 17. PMID 25044079